CLINICAL TRIAL: NCT03184155
Title: Prevention of Coronary Microvascular Dysfunction Post-PCI by Intracoronary Nicardipine
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: This study was planned, but recruitment and enrollment never began.
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 17D.172
Record Dates: First submitted 2017-06-07; First posted 2017-06-12 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease
Keywords: Nicardipine; Percutaneous Coronary Intervention; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Nicardipine

STUDY DESIGN:
Intervention Model Description: Randomized double blind, placebo controlled, study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intracoronary Nicardipine (Experimental): 200 mcg intracoronary injection of nicardipine prior to PCI, with potential for additional 100 mcg nicardipine before stent placement, balloon post-dilation, and before post-PCI IMR measurement.
  Interventions: Drug: Nicardipine
- Sterile Saline (Placebo Comparator): Injection of sterile saline prior to PCI, with potential for additional saline injections before stent placement, balloon post-dilation, and before post-PCI IMR measurement.
  Interventions: Drug: Sterile Saline

INTERVENTIONS:
Drug: Nicardipine — 200 mcg intracoronary nicardipine injection prior to PCI followed by an additional 2-4 doses of 100 mcg intracoronary nicardipine depending on complexity of PCI
  Arms: Intracoronary Nicardipine
Drug: Sterile Saline — Bolus of intracoronary sterile saline injection prior to PCI followed by an additional 2-4 doses of sterile saline depending on complexity of PCI
  Arms: Sterile Saline

SUMMARY:
This is a single-center double blind, placebo controlled study of patients undergoing a cardiac catheterization where the need for a percutaneous coronary intervention (PCI) is anticipated or will be determined during the early diagnostic phase. The study will assess the use of intracoronary nicardipine vs. sterile saline injection in reducing the index measurement of microcirculatory resistance (IMR). Fifty consecutive patients presenting to the Thomas Jefferson University (TJUH) Cardiac Catheterization lab will be randomized in a 1:1 fashion to receive either intracoronary nicardipine or sterile saline injection prior to PCI. IMR values will be assessed pre and post procedure. Data on clinical outcomes and adverse events will be collected by phone at 30 days and 1 year following the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Consenting adults age > 18 years
* Patients with stable coronary disease, stable angina, and/or objective evidence of myocardial ischemia OR
* Target vessel lesion with > 50% stenosis treated by PCI

Exclusion Criteria:

* Patients presenting with ST elevation myocardial infarction
* Complete total occlusion of the vessel
* Unprotected left main disease
* Presentation with acute coronary syndrome and actively rising troponin
* Contraindication to adenosine (advanced heart blocks, bronchospasm, HSN to the drug)
* Known hypersensitivity to nicardipine
* Severe aortic stenosis
* Left Ventricular dysfunction with ejection fraction less than 30%
* Hemodynamically unstable defined as systolic blood pressure < 90 mmHg and not responding to IV fluids
* Significant chronic renal insufficiency (Glomerular filtration rate [GFR] <30)
* Unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in Index of Microcirculatory Resistance (IMR) | From the start of the PCI procedure to immediately following the PCI procedure
  IMR is an intracoronary artery pressure measurement obtained during cardiac catheterization, and is a reliable indicator of microvascular dysfunction

SECONDARY OUTCOMES:
Post-Procedure myocardial Infarction (PMI) | 6-8 hours post procedure
  PMI is diagnosed by elevation of serum Troponin, 5 times the upper limit following a procedure.
Post-Procedure myocardial Infarction (PMI) | 12-18 hours post procedure
  PMI is diagnosed by elevation of serum Troponin, 5 times the upper limit following a procedure.
Major Adverse Cardiac Event | 30 Days following procedure
  Incidence of myocardial infarction, rehospitalization, or mortality
Major Adverse Cardiac Event | I year following procedure
  Incidence of myocardial infarction, rehospitalization, or mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michael Savage, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No